CLINICAL TRIAL: NCT02987322
Title: Honey Supplementation in Children With Idiopathic Dilated Cardiomyopathy: A Randomized Controlled Study
Brief Title: Honey in Idiopathic Dilated Cardiomyopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: mamdouh abdulmaksoud abdulrhman (Other)
Responsible Party: Sponsor-Investigator, mamdouh abdulmaksoud abdulrhman, professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4472/28.9.2015
Record Dates: First submitted 2016-11-29; First posted 2016-12-08 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Idiopathic Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Honey

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- honey (Experimental): Ziziphus honey (sider honey) orally in a dose of 1ml (1.2g)/kg/day for 3 months for the patients in the honey group.
  Interventions: Dietary Supplement: honey

INTERVENTIONS:
Dietary Supplement: honey — Ziziphus honey (sider honey) orally in a dose of 1ml (1.2g)/kg/day for 3 months

SUMMARY:
Background: Honey, as a natural product produced by honey bees, has anti-oxidant, anti-microbial, anti-inflammatory and immunomodulator properties. A few reports suggest that honey might have positive effects on cardiovascular diseases.

Methods: This was a randomized controlled study, which was carried out on 50 children, aged 2 to 12 years, suffering from idiopathic dilated cardiomyopathy (IDC). Patients were randomly assigned into two equal groups: the honey group and the control group. In the honey group, honey was provided in a dose of 1.2g/kg/day for three months in addition to the traditional treatment of IDC. The patients in the control group received only their standard treatment, without honey. The main outcome measure was the percent change in the ejection fraction (EF) and the fraction shortening (FS) shown in echocardiography.

DETAILED DESCRIPTION:
Background: Honey, as a natural product produced by honey bees, has anti-oxidant, anti-microbial, anti-inflammatory and immunomodulator properties. A few reports suggest that honey might have positive effects on cardiovascular diseases.

Methods: This was a randomized controlled study, which was carried out on 50 children, aged 2 to 12 years, suffering from idiopathic dilated cardiomyopathy (IDC). Patients were randomly assigned into two equal groups: the honey group and the control group. In the honey group, honey was provided in a dose of 1.2g/kg/day for three months in addition to the traditional treatment of IDC. The patients in the control group received only their standard treatment, without honey. The main outcome measure was the percent change in the ejection fraction (EF) and the fraction shortening (FS) shown in echocardiography. Patients in each group were subjected to history taking, clinical examination and investigations, including ECG and echocardiography at baseline and end of the study. Patients continued their standard treatment during the study. The honey used in the study was subjected to physicochemical analysis before use, and it was kept in closed containers away from light until the time of administration.

ELIGIBILITY:
Inclusion Criteria:

1. Echocardiographic diagnosis of dilated cardiomyopathy (DCM), based on the presence of left ventricular enlargement and systolic dysfunction with an ejection fraction <45%.
2. The echocardiographic findings included left ventricular dilatation and systolic dysfunction, with or without mitral regurgitation

Exclusion Criteria:

1. Other types of cardiomyopathy
2. Systemic or chronic illness, including cancer, endocrine disorders and sepsis
3. Children with diabetes mellitus
4. Ischemic heart disease diagnosed by coronary angiography or a history of myocardial infarction
5. Systemic hypertension with a blood pressure >170/100 mm Hg -

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Ejection fraction % as measured by echocardiography | 3 months
  The main outcome measure is the average increase or decrease of the ejection fraction (expressed as percentage), which refers to the amount, or percentage, of blood that is pumped (or ejected) out of the ventricles with each contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Elgendy, Lecturer, Principal Investigator — Ain Shams University, Pediatric departement

IPD SHARING:
Plan to Share IPD: Undecided
honey as a complementary or alternative treatment in cardiovascular diseases